CLINICAL TRIAL: NCT04735016
Title: DiamondTemp Global Registry
Status: Recruiting | Type: Observational
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT20059
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Treatment Arm: Patients enrolled and treated with the DiamondTemp™ Ablation System
  Interventions: Device: DiamondTemp™ Ablation System

INTERVENTIONS:
Device: DiamondTemp™ Ablation System — A cardiac ablation will be performed using the DiamondTemp™ Ablation System.

SUMMARY:
The DiamondTemp™ Global Registry is a prospective, global, multi-center, observational post-market registry.

DETAILED DESCRIPTION:
The DiamondTemp™ Global Registry is a prospective, global, multi-center, observational post-market registry. The purpose of this clinical study is to describe clinical performance and safety data in a broad patient population treated with the commercially available DiamondTemp™ Family of Cardiac Ablation Catheters (hereafter referred to as the DiamondTemp™ Ablation System) and followed according to the standard of care at each respective institution. The follow up period is intended to align with standard practice and subjects will be followed for a minimum of 12 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age or minimum age as required by local regulations
* Planned procedure using commercially available DiamondTemp™ Ablation System
* Willing to comply with study requirements and give IC (defined as legally effective, documented confirmation of a subject's voluntary agreement to participate in this clinical study) or authorization per institution and geographical requirements

Exclusion Criteria:

* Subject is enrolled in a concurrent study that has not been approved for concurrent enrollment by the global study manager
* Subject with exclusion criteria required by local law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects ≥ 18 years of age (or minimum age as required by local regulations) who have a recommendation for an ablation with the DiamondTemp™ Ablation System may be approached regarding enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Freedom from Recurrence at 12 Months | 12 Months
  Estimate the 12-month freedom from recurrence of the arrhythmia(s) treated at the study index ablation procedure using the DiamondTemp™ Ablation System.
Freedom from Device / Procedure Related Adverse Events | 12 Months
  Estimate serious device and serious procedure-related adverse events for ablation using the DiamondTemp™ Ablation System through 12 months.

CONTACTS AND LOCATIONS:
Locations (21):
- Australia (2):
  - Sunshine Coast University Hospital, Birtinya
  - Fiona Stanley Hospital, Murdoch
- Universitair Ziekenhuis Brussel, Jette, Belgium
- France (2):
  - CHRU de Tours - Hôpital Trousseau, Chambray-lès-Tours
  - Capio - Clinique du Tonkin, Villeurbanne
- Germany (3):
  - Herz- und Diabeteszentrum NRW - Ruhr-Universität Bochum, Bad Oeynhausen
  - Universitäres Herzzentrum, Hamburg
  - Saint Vincenz Krankenhaus Paderborn, Paderborn
- Italy (3):
  - Humanitas Mater Domini, Castellanza
  - Ospedale di Conegliano - S. Maria dei Battuti, Conegliano
  - Ospedale dell'Angelo, Venezia
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
- John Paul II Upper Silesian Medical Centre, Katowice, Poland
- Hospital de Santa Marta, Lisbon, Portugal
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- Spain (2):
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Inselspital - Universitätsspital Bern, Bern, Switzerland
- United Kingdom (2):
  - Royal Sussex County Hospital, Brighton
  - University Hospitals Coventry & Warwickshire, Coventry